CLINICAL TRIAL: NCT04343456
Title: Analysis of Benefit From Salvage Surgery for Highly Selected Patients With Metastatic Gastrointestinal Stromal Tumors Receiving Regorafenib Facing Local Progression
Brief Title: Salvage Surgery for Patients With Metastatic GIST With Rego
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chun-Nan Yeh, Principal investigator, Head of General Surgery, and Professor of Surgery, Chang Gung Memorial Hospital
Other Study IDs: Rego_op
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Gastrointestinal Stromal Tumors; Metastasis; Disease Progression
Keywords: regorafenib; Gastrointestinal Stromal Tumors; Metastasis; local progression; surgery
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis; Disease Progression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Salvage surgery with massive debulking — For patients with regorafenib treatment and facing local progression, we remove the tumor with progression and achieve cytoreduction.

SUMMARY:
Some researches have shown surgery may acquire progression-free (PFS) benefit for selected patients with metastatic gastrointestinal stromal tumor (GIST) who received first-line imatinib and second-line sunitinib. However, impact of salvage surgery on pre-treated GIST patients receiving third-line regorafenib facing progression is not yet reported. Investigators retrospectively reviewed patients with regorafenib treatment with salvage surgery.

DETAILED DESCRIPTION:
Between 2014 and 2019, 41 metastatic GIST patients received regorafenib therapy. 35 out of 41 metastatic GIST patients who were on regorafenib therapy facing progression and 15 experienced local progression underwent salvage surgery. Thirty-five of 41 (85.4 %) pre-treated GIST patients receiving regorafenib who experienced disease progression after a median follow-up of 12.4 months of regorafenib use. 15 out of 35 (42.9%) metastatic GIST patients receiving regorafenib facing progression underwent salvage surgery.

ELIGIBILITY:
Inclusion criteria:

1. Patients who is taking regorafenib after treatment failure by 1st line and 2nd line tyrosine kinase, namely Imatinib and Sunitinib.
2. Patients with aforementioned condition and is facing local progression of disease or stationary disease.

Exclusion criteria

1. Systemic progression of disease
2. ASA classification > 3

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between 2014 and 2019, 41 metastatic GIST patients receiving regorafenib therap at Chang Gung Memorial Hospital, Linkou, Taiwan were enrolled. All the patients were managed by a multidisciplinary GIST team composed of medical oncologists and surgical oncologists.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Overall survival | 01/2014~12/2019
  the time period from start regorafenib to death
Disease free survival | 01/2014~12/2019
  the time period after salvage surgery to disease reprogression

CONTACTS AND LOCATIONS:
Overall Officials: Chun Nan Yeh, MD., Study Director — Chang Gung Memorial Hospital, Linkuo
Locations (1):
- Chang Gung Memorial Hospital Linkou Branch, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No